CLINICAL TRIAL: NCT01143246
Title: A Multi-Center, Randomized, Placebo-controlled, Double-Blind Study to Confirm the Reversal of Hepatorenal Syndrome Type 1 With Lucassin® (Terlipressin) (The REVERSE Study)
Brief Title: A Placebo-Controlled, Double-Blind Study to Confirm the Reversal of Hepatorenal Syndrome Type 1 With Terlipressin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IK-4001-HRS-301
Record Dates: First submitted 2010-06-11; First posted 2010-06-14 (Estimated); Results first posted 2022-11-29 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Hepatorenal Syndrome
Keywords: Hepatorenal syndrome; Renal failure; Cirrhosis; Alcoholic hepatitis; Ascites
MeSH Terms: conditions — Hepatorenal Syndrome; Renal Insufficiency; Fibrosis; Hepatitis, Alcoholic; Ascites | interventions — Terlipressin; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Terlipressin (Experimental): Participants receive terlipressin intravenously as a bolus injection, followed by a saline flush. Dose, duration, retreatment and/or discontinuation may be modified by the investigator, per protocol.
  Interventions: Drug: Terlipressin
- Placebo (Placebo Comparator): Participants receive matching placebo intravenously as a bolus injection, followed by a saline flush. Dose, duration, retreatment and/or discontinuation may be modified by the investigator, per protocol.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Terlipressin — Each 6 mL vial contains 1 mg lyophilized terlipressin acetate and 10 mg mannitol in sterile 0.9% sodium chloride solution.
  Other Names: Lucassin®
  Arms: Terlipressin
Drug: Placebo — 11 mg mannitol reconstituted with 5 ml of sterile 0.9% sodium chloride solution.
  Other Names: Saline
  Arms: Placebo

SUMMARY:
This study is designed to evaluate the efficacy and safety of intravenous terlipressin versus placebo for the treatment of type 1 hepatorenal syndrome (HRS) in participants receiving standard of care albumin therapy.

DETAILED DESCRIPTION:
Hepatorenal syndrome is a rare syndrome of marked renal dysfunction in patients with cirrhosis, decompensated liver disease, and portal hypertension. Hepatorenal syndrome type 1 is characterized by a rapid progressive renal impairment and has a very poor prognosis with > 80% mortality within 3 months. At present, there are no approved drug therapies for HRS type 1 in the US, Australia, or Canada. The only curative treatment for HRS type 1 and the underlying end-stage cirrhosis is liver transplantation. However, many patients will not survive long enough to receive a liver transplant and therapy, which may provide a bridge to transplantation, is badly needed. Increased understanding of the pathophysiology of HRS type 1 has demonstrated that vasoconstrictive drug therapy may reverse HRS type 1. Substantial data available from many published clinical investigations in the literature provide compelling evidence suggesting that administration of terlipressin improves renal function in patients with HRS.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent by subject or legally authorized representative
2. At least 18 years of age
3. Cirrhosis and ascites
4. Rapidly progressive reduction in renal function characterized by:

   * Serum creatinine (SCr) ≥ 2.5 mg/dL
   * Doubling of SCr within 2 weeks (or for observations of shorter duration, SCr values over time meeting slope-based criteria for proportional increases likely to be representative of at least a doubling within 2 weeks
5. No sustained improvement in renal function (< 20% decrease in SCr and SCr ≥ 2.25 mg/dL) 48 hours after both diuretic withdrawal and the beginning of plasma volume expansion with albumin:

Note: Albumin doses recommended by the International Ascites Club (IAC) are 1 g/kg on the first day (Maximum 100 g) and 20 - 40 g/day thereafter as clinically indicated. It is recommended (if clinically appropriate) that the albumin dose is kept constant during the study drug administration period.

Note: The qualifying SCr value is the SCr value at least 48 hrs after both diuretic withdrawal (if applicable) and the beginning of albumin fluid challenge. The qualifying SCr value must be ≥ 2.25 mg/dL AND at least 80% of the diagnostic (pre-fluid challenge) SCr value.

Exclusion Criteria:

1. SCr > 7 mg/dL
2. Shock Note: Hypotension (Mean Arterial Pressure < 70 mm Hg or a decrease > 40 mm Hg in systolic blood pressure from baseline) with evidence of hypoperfusion abnormalities despite adequate fluid resuscitation.
3. Sepsis or systemic inflammatory response syndrome (SIRS)

   Note: SIRS: Presence of 2 or more of the following findings:

   Temperature > 38°C or < 36°C; heart rate > 90/min; respiratory rate of > 20/min or a PaCO2 of < 32 mm Hg; white blood cell count of > 12,000 cells/µL or < 4,000/ µL.

   Note: Sepsis: Documented infection and systemic inflammatory response syndrome.
4. < 2 days anti-infective therapy for documented or suspected infection
5. Proteinuria > 500 mg/day
6. Hematuria or microhematuria (> 50 red blood cells per high power field)
7. Clinically significant casts on urinalysis, including granular casts Note: Urine sediment examination is required to exclude presence of granular casts and other clinically significant casts [e.g., red blood cell (RBC) casts].
8. Evidence of intrinsic or parenchymal renal disease (including acute tubular necrosis)
9. Obstructive uropathy or other renal pathology on ultrasound or other medical imaging
10. Current or recent treatment (within 4 weeks) with nephrotoxic drugs, e.g., aminoglycosides, nonsteroidal anti-inflammatory drugs (NSAID) Note: Up to 3 doses of an NSAID within the prior month (prescription or over the counter) is acceptable Note: Use of short-term (< 2 weeks) oral neomycin for acute encephalopathy is acceptable.
11. Current or recent (within 4 weeks) renal replacement therapy
12. Superimposed acute liver failure/injury due to factors other than alcoholic hepatitis, including acute viral hepatitis, drugs, medications (e.g., acetaminophen), or other toxins (e.g., mushroom [Amanita] poisoning)
13. Current or recent treatment (within 48 hours) with octreotide, midodrine, vasopressin, dopamine or other vasopressors
14. Severe cardiovascular disease as judged by investigator
15. Estimated life expectancy of less than 3 days
16. Confirmed pregnancy
17. Known allergy or sensitivity to terlipressin or another component of the study treatment
18. Participation in other clinical research studies involving the evaluation of other investigational drugs or devices within 30 days of randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2010-10-11 (Actual); Primary Completion 2013-02 (Actual); Study Completion 2013-05-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Team Leader, Study Director — Mallinckrodt
Locations (73):
- United States (71):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Banner Good Samaritan Medical Center/Liver Disease Center, Phoenix, Arizona
  - Mayo Clinic Arizona, Phoenix, Arizona
  - University of Arizona Medical Center South Campus, Tucson, Arizona
  - University of Arizona Liver Research Institute, Tucson, Arizona
  - Arrowhead Regional Medical Center, Colton, California
  - SCTI Research Foundation, Coronado, California
  - Scripps Clinic, La Jolla, California
  - USC University Hospital, Los Angeles, California
  - UC Davis Medical Center, Sacramento, California
  - Veteran's Administration Medical Center, San Diego, California
  - California Pacific Medical Center, San Francisco, California
  - University of Colorado Denver, Aurora, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Yale University School of Medicine, New Haven, Connecticut
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - Mayo Clinic, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Indiana University Health - University Hospital, Indianapolis, Indiana
  - Iowa City VA Health Care System, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - University of Louisville, Louisville, Kentucky
  - Tulane Medical Center, New Orleans, Louisiana
  - University of Maryland, Baltimore, Maryland
  - Beth Lsrael Deaconess Medical Center, Boston, Massachusetts
  - Lahey Clinic Medical Center, Burlington, Massachusetts
  - University of Massachusetts Medical Center, Worcester, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Saint Luke's Hospital, Kansas City, Missouri
  - Saint Louis University, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Bellevue Hospital, New York, New York
  - NYU Langhorn Medical Center, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - New York Medical College/Westchester Medical Center, Valhalla, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - University of Cincinnati, Internal Medicine-Digestive Diseases, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - INTEGRIS Baptist Medical Center, Oklahoma City, Oklahoma
  - Orgeon Health & Science University, Portland, Oregon
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania
  - VA Pittsburgh Healthcare System, Pittsburgh, Pennsylvania
  - WJB Dorn VA Medical Center, Columbia, South Carolina
  - Vanderbilt Medical Center, Nashville, Tennessee
  - Dallas VA Medical Center, Dallas, Texas
  - Baylor University Medical Center, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Baylor All Saints Medical Center, Fort Worth, Texas
  - The University of Texas Medical Branch at Galveston, Galveston, Texas
  - St. Luke's Advanced Liver Therapies, Houston, Texas
  - The Methodist Hospital, Houston, Texas
  - University of Texas Health Science Center at Houston - Memorial Hermann Hospital, Houston, Texas
  - Methodist Specialty Transplant Hospital Lab, San Antonio, Texas
  - The University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University of Texas Health Science Center, San Antonio, Texas
  - University of Utah, Salt Lake City, Utah
  - McGuire DVAMC, Richmond, Virginia
  - Virginia Commonwealth University Health System, Richmond, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin
- Canada (2):
  - Toronto General Hospital, Toronto, Ontario
  - CHUM, Hopital St-Luc, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No
Discussion of statistical endpoints and analysis are included in manuscripts. Summary aggregate (basic) results (including adverse events information) and the study protocol are made available on clinicaltrials.gov (NCT02770716) when required by regulation. Individual de-identified patient data will not be disclosed. Requests for additional information should be directed to the company at medinfo@mnk.com.

REFERENCES:
- [Derived] Bajaj JS, Kwo P, Pappas SC, O'Leary JG, Jamil K, Cardoza S, Wong F. Bradycardia and Other Arrhythmias in Patients With Hepatorenal Syndrome-Acute Kidney Injury Following Terlipressin Treatment: A Pooled Analysis of Three North American Phase III Clinical Studies. Aliment Pharmacol Ther. 2025 Dec;62(11-12):1192-1201. doi: 10.1111/apt.70297. Epub 2025 Jul 24. PMID 40704461
- [Derived] Mujtaba MA, Gamilla-Crudo AK, Merwat SN, Hussain SA, Kueht M, Karim A, Khattak MW, Rooney PJ, Jamil K. Terlipressin in combination with albumin as a therapy for hepatorenal syndrome in patients aged 65 years or older. Ann Hepatol. 2023 Sep-Oct;28(5):101126. doi: 10.1016/j.aohep.2023.101126. Epub 2023 Jun 10. PMID 37302573
- [Derived] Velez JCQ, Wong F, Reddy KR, Sanyal AJ, Vargas HE, Curry MP, Gonzalez SA, Pappas SC, Jamil K. The Effect of Terlipressin on Renal Replacement Therapy in Patients with Hepatorenal Syndrome. Kidney360. 2023 Aug 1;4(8):1030-1038. doi: 10.34067/KID.0000000000000132. Epub 2023 May 5. PMID 37143199
- [Derived] Curry MP, Vargas HE, Befeler AS, Pyrsopoulos NT, Patwardhan VR, Jamil K. Early treatment with terlipressin in patients with hepatorenal syndrome yields improved clinical outcomes in North American studies. Hepatol Commun. 2023 Jan 3;7(1):e1307. doi: 10.1097/01.HC9.0000897228.91307.0c. eCollection 2023 Jan 1. PMID 36633470
- [Derived] Sanyal AJ, Boyer TD, Frederick RT, Wong F, Rossaro L, Araya V, Vargas HE, Reddy KR, Pappas SC, Teuber P, Escalante S, Jamil K. Reversal of hepatorenal syndrome type 1 with terlipressin plus albumin vs. placebo plus albumin in a pooled analysis of the OT-0401 and REVERSE randomised clinical studies. Aliment Pharmacol Ther. 2017 Jun;45(11):1390-1402. doi: 10.1111/apt.14052. Epub 2017 Mar 29. PMID 28370090
- [Derived] Wong F, Pappas SC, Boyer TD, Sanyal AJ, Bajaj JS, Escalante S, Jamil K; REVERSE Investigators. Terlipressin Improves Renal Function and Reverses Hepatorenal Syndrome in Patients With Systemic Inflammatory Response Syndrome. Clin Gastroenterol Hepatol. 2017 Feb;15(2):266-272.e1. doi: 10.1016/j.cgh.2016.07.016. Epub 2016 Jul 25. PMID 27464593
- [Derived] Boyer TD, Sanyal AJ, Wong F, Frederick RT, Lake JR, O'Leary JG, Ganger D, Jamil K, Pappas SC; REVERSE Study Investigators. Terlipressin Plus Albumin Is More Effective Than Albumin Alone in Improving Renal Function in Patients With Cirrhosis and Hepatorenal Syndrome Type 1. Gastroenterology. 2016 Jun;150(7):1579-1589.e2. doi: 10.1053/j.gastro.2016.02.026. Epub 2016 Feb 16. PMID 26896734

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 52 active sites in the United States and Canada.
Period: Overall Study
Arm/Group | Terlipressin | Placebo
Started | 97 | 99
Intent to Treat (ITT) (All randomized participants who had at least one baseline assessment.) | 97 | 99
Safety Population (Treated Participants) (Eight participants did not receive treatment and were excluded from Safety Population.) | 93 | 95
Completed | 52 | 48
Not Completed | 45 | 51
Not completed — Adverse Event | 24 | 28
Not completed — Participant Withdrew Informed Consent | 2 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Death | 16 | 15
Not completed — Reason not Specified | 3 | 5

BASELINE CHARACTERISTICS:
Population: ITT population.
Groups:
- Terlipressin; Placebo: Participants receive matching placebo intravenously as a bolus injection, followed by a saline flush. Dose, duration, retreatment and/or discontinuation may be modified by the investigator, per protocol.
- Total: Total of all reporting groups
Arm/Group | Terlipressin | Placebo | Total
Number analyzed (Participants) | 97 | 99 | 196
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.8 (8.38) | 54.8 (8.50) | 55.3 (8.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 32 | 77
  Male | 52 | 67 | 119
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 15 | 25
  Not Hispanic or Latino | 86 | 84 | 170
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 6 | 13
  White | 85 | 92 | 177
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Canada | 5 | 4 | 9
  United States | 92 | 95 | 187

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Confirmed Hepatorenal Syndrome (HRS) Reversal
Description: Confirmed HRS Reversal: The percentage of participants with two serum creatinine (SCr) values of ≤ 1.5 mg/dL at least 48 hours apart, on treatment, and without intervening renal replacement therapy or liver transplant.
Time Frame: within 14 days
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Terlipressin | Placebo
Number analyzed (Participants) | 97 | 99
percentage of participants | 19.6 | 13.1

2. Secondary Outcome: Percentage of Participants With HRS Reversal
Description: HRS reversal is defined as at least one SCr value of ≤ 1.5 mg/dL on treatment (up to 24 hours after the last dose of study medication).
Time Frame: within 14 days
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Terlipressin | Placebo
Number analyzed (Participants) | 97 | 99
percentage of participants | 23.7 | 15.2

3. Secondary Outcome: Percentage of Participants With Transplant-free Survival
Description: Transplant-Free Survival up to 90 days, defined as the time (in days) that each participant survives without liver transplantation from the day of randomization.
Time Frame: Up to 90 days
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Terlipressin | Placebo
Number analyzed (Participants) | 97 | 99
percentage of participants | 30.9 | 26.3

4. Secondary Outcome: Percentage of Participants With Overall Survival
Description: Overall Survival up to 90 days, defined as the time (in days) that each participant survives from the day of randomization.
Time Frame: Up to 90 days
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Terlipressin | Placebo
Number analyzed (Participants) | 97 | 99
percentage of participants | 57.7 | 54.5

5. Secondary Outcome: Percentage of Participants With Serious Adverse Events
Description: Clinically significant changes in vital signs, height, weight, immunogenicity and laboratory assessments which qualified for the definition of serious adverse event are reported.
Time Frame: Up to 30 days post treatment (within 44 days)
Population: Safety population.
Measure: Number; unit: percentage of participants
Arm/Group | Terlipressin | Placebo
Number analyzed (Participants) | 93 | 95
percentage of participants | 66.7 | 62.1

ADVERSE EVENTS:
Time Frame: All-cause mortality was reported for the ITT population. SAEs are collected in the safety analysis set (SAS) from informed consent to 30 days post-treatment (up to approximately 44 days); deaths are collected through study completion at 90 days from treatment start. Other adverse events were collected up to 7 days of treatment.
Description: Participants experiencing multiple episodes of a given adverse event are counted once within each preferred term and within each system organ class in the Safety population.
Arm/Group | Terlipressin | Placebo
All-Cause Mortality (participants affected / at risk) | 41/97 | 45/99
Serious Adverse Events (participants affected / at risk) | 62/93 | 59/95
Other Adverse Events (participants affected / at risk) | 87/93 | 82/95
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Terlipressin (N=93) | Placebo (N=95)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 0 (0) | 4 (4)
Cardiac Failure Congestive (Cardiac disorders) | 1 (1) | 0 (0)
Cardio-Respiratory Arrest (Cardiac disorders) | 2 (2) | 1 (1)
Cardiogenic Shock (Cardiac disorders) | 1 (1) | 0 (0)
Cyanosis (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial Ischaemia (Cardiac disorders) | 0 (0) | 1 (1)
Stress Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Tachyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal Compartment Syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 5 (7) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 3 (3)
Colitis Ischaemic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1)
Ileus Paralytic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal Ischaemia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Intra-abdominal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal Perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal Varices Haemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1)
Pancreatitis Acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 2 (2) | 1 (1)
Cardiac Death (General disorders) | 0 (0) | 1 (1)
Chest Pain (General disorders) | 0 (0) | 1 (1)
Multiple Organ Dysfunction Syndrome (General disorders) | 12 (12) | 6 (6)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Bile Duct Necrosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Chronic Hepatic Failure (Hepatobiliary disorders) | 9 (10) | 8 (8)
Cirrhosis Alcoholic (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hepatic Artery Thrombosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic Cirrhosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic Failure (Hepatobiliary disorders) | 4 (4) | 6 (6)
Hepatorenal Failure (Hepatobiliary disorders) | 2 (2) | 1 (1)
Hepatorenal Syndrome (Hepatobiliary disorders) | 7 (7) | 2 (2)
Liver Transplant Rejection (Immune system disorders) | 0 (0) | 1 (1)
Abdominal Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 1 (2)
Clostridium Difficile Colitis (Infections and infestations) | 1 (1) | 0 (0)
Enterococcal Infection (Infections and infestations) | 2 (2) | 0 (0)
Mediastinitis (Infections and infestations) | 0 (0) | 1 (1)
Peritonitis Bacterial (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 5 (5)
Sepsis (Infections and infestations) | 4 (4) | 3 (3)
Septic Shock (Infections and infestations) | 4 (4) | 2 (2)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 1 (1)
Urinary Tract Infection Fungal (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Hepatic Haematoma (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hip Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post Procedural Bile Leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural Haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 2 (3)
Toxicity To Various Agents (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Transfusion-Related Acute Lung Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Transplant Failure (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood Creatinine Increased (Investigations) | 1 (1) | 1 (1)
Blood Urea Increased (Investigations) | 0 (0) | 1 (1)
White Blood Cell Count Increased (Investigations) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Metabolic Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hepatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhage Intracranial (Nervous system disorders) | 0 (0) | 1 (1)
Hepatic Encephalopathy (Nervous system disorders) | 1 (1) | 3 (3)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Subarachnoid Haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Mental Status Changes (Psychiatric disorders) | 1 (1) | 1 (1)
Renal Failure (Renal and urinary disorders) | 3 (4) | 4 (4)
Renal Impairment (Renal and urinary disorders) | 3 (3) | 0 (0)
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Obstructive Airways Disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Respiratory Arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 1 (1)
Vascular Skin Disorder (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Withdrawal Of Life Support (Surgical and medical procedures) | 0 (0) | 1 (1)
Haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 2 (2) | 4 (4)
Hypovolaemic Shock (Vascular disorders) | 1 (1) | 0 (0)
Poor Peripheral Circulation (Vascular disorders) | 1 (1) | 0 (0)
Oliguria (Renal and urinary disorders) | 2 (2) | 0 (0)
Death (General disorders) | 1 (1) | 1 (1)
Liver disorder (Hepatobiliary disorders) | 1 (1) | 0 (0)
Klebsiella sepsis (Infections and infestations) | 1 (1) | 0 (0)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 2 (3)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Terlipressin (N=93) | Placebo (N=95)
Anaemia (Blood and lymphatic system disorders) | 10 (10) | 9 (10)
Coagulopathy (Blood and lymphatic system disorders) | 5 (5) | 4 (4)
Bradycardia (Cardiac disorders) | 9 (10) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 6 (6) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 26 (27) | 21 (22)
Diarrhoea (Gastrointestinal disorders) | 22 (22) | 4 (4)
Nausea (Gastrointestinal disorders) | 12 (12) | 12 (12)
Vomiting (Gastrointestinal disorders) | 9 (9) | 5 (5)
Oedema peripheral (General disorders) | 6 (7) | 8 (9)
Pyrexia (General disorders) | 6 (6) | 5 (5)
Hepatorenal syndrome (Hepatobiliary disorders) | 2 (2) | 9 (9)
Urinary tract infection (Infections and infestations) | 4 (4) | 6 (6)
Fluid overload (Metabolism and nutrition disorders) | 9 (9) | 5 (5)
Hyperglycaemia (Metabolism and nutrition disorders) | 6 (6) | 2 (2)
Hyperphosphataemia (Metabolism and nutrition disorders) | 5 (5) | 5 (5)
Hypokalaemia (Metabolism and nutrition disorders) | 11 (11) | 5 (5)
Hypophosphataemia (Metabolism and nutrition disorders) | 5 (5) | 2 (2)
Metabolic acidosis (Metabolism and nutrition disorders) | 10 (10) | 7 (7)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6 (7) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1)
Asterixis (Nervous system disorders) | 8 (8) | 4 (4)
Headache (Nervous system disorders) | 6 (6) | 5 (5)
Hepatic encephalopathy (Nervous system disorders) | 8 (8) | 11 (11)
Lethargy (Nervous system disorders) | 9 (9) | 3 (3)
Anxiety (Psychiatric disorders) | 6 (8) | 3 (3)
Insomnia (Psychiatric disorders) | 6 (6) | 3 (3)
Mental status changes (Psychiatric disorders) | 5 (5) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 8 (9)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 5 (5)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 4 (6)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 5 (5)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 6 (6) | 3 (3)
Hypotension (Vascular disorders) | 17 (18) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Disclosure of individual investigator/site results is restricted for 18 months after final evaluation of study results or after release of a cooperative publication including all study from all sites, whichever occurs first. The sponsor has 60 days to review and comment on the publication and can request removal of any confidential information prior to public disclosure or publication.